CLINICAL TRIAL: NCT04832763
Title: Colorectal Cancer in Adolescents and Young Adults: A Pilot Study of Medical and Psychosocial Issues
Brief Title: Medical and Psychosocial Issues in Adolescents and Young Adults With Colorectal Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3C-19-4; NCI-2020-02581 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 3C-19-4 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2020-05-09; First posted 2021-04-06 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Stage I Colorectal Cancer AJCC v8; Stage II Colorectal Cancer AJCC v8; Stage IIA Colorectal Cancer AJCC v8; Stage IIB Colorectal Cancer AJCC v8; Stage IIC Colorectal Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Physical function testing, questionnaire (Experimental): Patients on active treatment complete questionnaires and undergo collection of blood samples and physical function assessments at baseline, and at 3 and 6 months. Survivors in surveillance complete questionnaires and undergo collection of blood sample and physical function assessment at baseline.
  Interventions: Procedure: Biospecimen Collection; Other: Medical Chart Review; Other: Physical Performance Testing; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood sample
Other: Medical Chart Review — Review of medical charts
  Other Names: Chart Review
Other: Physical Performance Testing — Undergo physical function testing
  Other Names: Physical Fitness Testing; Physical Function Testing
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaire

SUMMARY:
This study investigates the medical and psychosocial consequences of colorectal cancer on adolescents and young adults. Measuring physical function in adolescents and young adults with colorectal cancer may help doctors better understand the level of physical function during cancer treatment and how to improve the management of colorectal cancer in adolescents and young adults. This study may also help design a future exercise program to decrease risk factors including high blood pressure, high blood sugar, and high cholesterol.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To prospectively characterize the symptom burden and assess the health-related quality of life of adolescents and young adults (AYAs) in active treatment for colorectal cancer in comparison to older patients to identify differences that contribute to the development of appropriately timed, age appropriate interventions.

II. To characterize the symptom burden and assess the health-related quality of life of AYAs who have completed curative therapy and are in surveillance for colorectal cancer compared to older patients to identify differences that contribute to the development of appropriately timed, age-appropriate interventions.

SECONDARY OBJECTIVE:

I. Using a prospective and cross-sectional design, characterize physical function, body composition, and biomarkers of comorbid conditions among AYAs with colorectal cancer (CRC) on active therapy and after completion of therapy in survivorship to identify targets for and timing of interventions.

EXPLORATORY OBJECTIVE:

I. To assess across Aims differences by cancer site (colon versus [vs.] rectal) by sex, and by race/ethnicity.

OUTLINE:

Patients on active treatment complete questionnaires and undergo collection of blood samples and physical function assessments at baseline, and at 3 and 6 months. Survivors in surveillance complete questionnaires and undergo collection of blood sample and physical function assessment at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of colorectal cancer (any stage)
* Any type of prior therapy
* Age >= 18-39 years for AYA/young adult sample, age 40+ for older comparison group
* For patients on active therapy: must have been diagnosed within the past three months. For survivors: must have completed curative therapy and are 6-24 months post-diagnosis
* Speak English or Spanish
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients who are more than 3 months from diagnosis, and survivors who are more than 24 months from initial diagnosis
* Patients who have a life expectancy of less than 6 months per their medical oncologist
* Patients who are deemed too ill or unable to participate by their medical oncologist (e.g., have cognitive impairment or brain metastases)
* Patients who do not speak English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptom Burden | Up to 6 months
  Symptom burden will be assessed with computer adaptive tests (CATs) from the PROMIS measurement system. PROMIS is an NIH-sponsored system for measuring patient-reported health status, including physical, mental, and social well-being. Participants will complete the PROMIS Anxiety, Depression, Fatigue, and Pain Interference computer adaptive tests (CATs), which administer the minimum number of items necessary to accurately measure patient-reported outcomes while minimizing participant burden.
Change in health-related quality of life (HRQoL) | Baseline up to 6 months
  HRQoL will be measured using the Functional Assessment of Cancer Therapy-Colorectal (FACT-C) Quality of Life Instrument, a disease-specific quality of life measure. The FACT-C includes 38 items assessing five domains of health-related quality of life: Physical, Social/Family, Emotional and Functional Well-Being, and a subscale that examines health symptoms specific to CRC patients. Participants evaluate how they have been feeling over the preceding week on a five-point Likert-type scale with a possible total score of 0 to 136, with higher scores reflecting better QoL.

SECONDARY OUTCOMES:
Physical function - cardiorespiratory fitness | Up to 6 months
  Physical function will be measured using the following in-lab test for cardiorespiratory fitness (6-minute walk test): 6-minute Walk Test (6MWT): Participants will be instructed to walk as quickly as possible without running on an indoor pre-measured walkway for 6 minutes. The investigator will follow behind the participant so as not to pace the participant, and record the distance covered. Approximate time: 10 minutes.
Physical function - power (stair climb) | Up to 6 months
  Functional power will be measured using a stair climb test (Margaria Stair Climb) that has been successfully performed and correlated with lower-extremity power and mobility performance in older adults with a reliability coefficient of 0.99. Participants will be instructed to ascend a flight of 10 stairs one step at a time as quickly as possible without using a handrail. Timing will begin when one foot steps on the 3rd stair, and ends when one foot reaches the 9th stair. Time is recorded to the nearest .01 second, and an average of 3 trials is calculated. One practice trial will be given before the 3 trials.
  Approximate time: 5 minutes.
Physical function - Mobility | Up to 6 months
  Mobility will be assessed using the Timed Up and Go (TUG) test, which has been shown to predict immediate fall risk better than static balance tests or isometric muscle strength. Participants begin seated in a chair with hands on the armrests, are asked to rise, walk to a line on the floor 3 meters from the chair, turn around, and return to the same seated position as quickly and safe as possible. Scores will be taken as the time to complete the task, with one practice trial given. An average of time for 3 trials is calculated. Approximate time: 5 minutes
Body composition | Up to 6 months
  Body composition will be assessed via bioelectrical impedance using a validated device (InBody 570, Cerritos, CA). Participants will be asked to remove their shoes and socks and stand still on the device while holding the handles with their hands at their sides. The device will estimate body fat using an algorithm based on their age, sex, height, and body weight. A tape measure will be used to obtain hip circumference defined as the distance around the widest girth of the buttocks using the greater trochanter as a landmark. A tape measure will be used to obtain waist circumference defined as the distance around the midpoint between the last palpable rib and top of the iliac crest.
Biomarker analysis - insulin | Up to 6 months
  Fasting insulin levels measured in blood
Biomarker analysis - glucose | Up to 6 months
  Fasting glucose levels measured in blood
Biomarker analysis - C-Reactive Protein | Up to 6 months
  C- reactive protein levels measured in blood

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Miller, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California